CLINICAL TRIAL: NCT06047821
Title: The Incidence and Burden of Shigella Diarrhea in Children Aged 6-35 Months: the Enterics for Global Health (EFGH) - Shigella Burden Study
Brief Title: Enterics for Global Health (EFGH)
Acronym: EFGH
Status: Active, not recruiting | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Aga Khan University (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); University of Maryland, Baltimore (Other); University of Virginia (Other); Asociacion Benefica Prisma (Other); Medical Research Council Unit, The Gambia (Other); Kenya Medical Research Institute (Other); Center for Vaccine Development - Mali (Other); Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Patricia B Pavlinac, Associate Professor, University of Washington
Other Study IDs: INV-01665
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Shigella; Child; Diarrhea
Keywords: Epidemiology; Shigella; Diarrhea; Children; Enterics; Vaccine
MeSH Terms: conditions — Dysentery, Bacillary; Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Shigella isolates, lactose fermenting sweep, and rectal swab/stool DNA; Specimens stored at -80 degrees Celsius at each respective country-site
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with Shigella Diarrhea: Children with Shigella identified by culture or quantitative PCR
- Children without Shigella Diarrhea: Children without Shigella identified by culture or quantitative PCR

SUMMARY:
Diarrhea remains a leading cause of death among young children, with the majority of diarrhea deaths occurring in low- and middle-income countries. Childhood diarrhea caused by a type of bacteria called "Shigella" is responsible for an estimated 60,000 deaths each year and may cause particularly severe illness among children. Currently, there are several promising vaccines to prevent Shigella diarrhea in development, but key information is still needed to inform future vaccine studies. The purpose of this study, titled Enterics for Global Health (or the "EFGH"), is to determine the number and rate of new cases of Shigella diarrhea among children 6 to 35 months of age presenting to health facilities with diarrhea or dysentery. Over a two-year period, the EFGH study will enroll 1,400 children from each of the seven countries: Peru, Pakistan, Bangladesh, Mali, Malawi, Kenya, and The Gambia (9,800 children total).

DETAILED DESCRIPTION:
In low- and middle-income countries, nearly one third of children experience at least one episode of Shigella-attributable diarrhea during their first 2 years of life. In addition to it being a leading cause of diarrhea, this enteric bacterium is also associated with linear growth faltering, a precursor to stunting. Stunting is a marker of vulnerability to childhood infection, decreased vaccine efficacy and lifelong morbidity. Currently, several promising Shigella vaccines are in development. Eventual Phase 2b/3 Shigella vaccine trials will require a consortium of potential vaccine trial sites in settings with a high incidence of Shigella-attributed medically-attended diarrhea, high participant retention, and the laboratory capacity to confirm Shigella infection. The Enterics for Global Health (EFGH) Shigella burden study will employ cross-sectional and longitudinal study designs to establish updated incidence rates and document consequences of Shigella diarrhea within 7 country sites in Africa, Asia, and Latin America. Over a two-year period, the EFGH study will enroll 9,800 children (1,400 per country site) between 6-35 months with medically-attended diarrhea. Through this multi-country surveillance network, selected EFGH sites will be ready to quickly implement rigorous and efficient vaccine trials and provide critical data to policy makers about the relative importance of this vaccine-preventable disease, accelerating the time to vaccine availability and uptake among children in high Shigella burden settings.

Primary Aims

1. Determine the incidence of Shigella-attributed medically-attended diarrhea in children 6 to 35 months of age in each of the EFGH country sites.

Secondary Aims

1. Determine the incidence of Shigella medically-attended diarrhea by serotype, severity definition, laboratory method (culture vs. qPCR), age, and by season.
2. Describe the prevalence of resistance to commonly used antibiotics in Shigella isolates in each EFGH country site.
3. Determine the risk of death, hospitalization, persistent diarrhea, diarrhea recurrence, and linear growth faltering in the 3 months following an episode of Shigella medically-attended diarrhea.
4. Compare various severity definitions in their ability to distinguish Shigella from non-Shigella attributable diarrhea and ability to predict risk of death or hospitalization in the subsequent 3 months.
5. Quantify the cost incurred by families and health care systems due to Shigella morbidity and mortality.
6. Identify optimal laboratory methods for Shigella culture by:

   1. comparing the isolation rate of Shigella between two transport media for rectal swabs (Cary-Blair and modified Buffered Glycerol Saline [BGS])
   2. comparing the isolation rate of Shigella between two fecal sample types (rectal swabs and whole stool) among the subset of children who produced whole stool in The Gambia and Bangladesh country sites.

ELIGIBILITY:
Inclusion Criteria:

1. Child is 6-35 months of age
2. Primary caregiver and child plan to remain at their current residence for at least the next 4 months
3. Primary caregiver is able to provide informed consent (legal age or emancipated minor) and provides consent within a common language for which translations are available
4. Child presents to health facility with diarrhea (≥3 abnormally loose or watery stools in the previous 24 hours) with or without the presence of blood
5. Child resides within the pre-defined study area
6. Fewer than 4 hours have passed since the child presented to a health facility
7. Diarrhea episode is:

   * Acute (onset within 7 days of study enrollment) and
   * Represents a new episode (onset after at least 2 diarrhea-free days)
8. Caregiver is willing to have child participate in follow-up visits at week 4 and month 3
9. Willingness to have samples collected from the child (rectal swabs at enrollment)
10. Site enrollment cap has not been met
11. Child is not being referred to a non-EFGH facility at the time of screening

Exclusion Criteria:

* Child is < 6-35 months of age
* Child is > 6-35 months of age
* Primary caregiver and child do not plan to remain at their current residence for at least the next 4 months
* Primary caregiver is not able to provide informed consent (legal age or emancipated minor)
* Primary caregiver does not provide consent within a common language for which translations are available
* Child does not present to health facility with diarrhea (≥3 abnormally loose or watery stools in the previous 24 hours) with or without the presence of blood
* Child does not reside within the pre-defined study area
* 4 or more hours have passed since the child presented to a health facility
* Diarrhea episode is not Acute (onset within 7 days of study enrollment)
* Diarrhea episode does not represent a new episode (onset after at least 2 diarrhea-free days)
* Caregiver is unwilling to have child participate in follow-up visits at week 4 and month 3
* Unwillingness to have samples collected from the child (rectal swabs at enrollment)
* Site enrollment cap has been met
* Child is being referred to a non-EFGH facility at the time of screening

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 6-35 months of age presenting with diarrhea at selected study health facilities in Bangladesh, Malawi, Kenya, Mali, the Gambia, Pakistan, and Peru.
Sampling Method: Non-Probability Sample
Enrollment: 9800 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2024-08-17 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Shigella incidence | At enrollment in the study (cross-sectional)
  The primary outcome measure is Shigella incidence, defined as incident diarrhea among children enrolled at health clinics attributable to Shigella by microbiological methods (culture or qPCR) divided by the estimated population living in the catchment area. Incidence will be reported as crude incidence as well as adjusted for healthcare seeking and the percentage of children who were enrolled.

SECONDARY OUTCOMES:
Antimicrobial susceptibility | At enrollment in the study (cross-sectional)
  Antimicrobial susceptibility will be computed separately for Ampicillin, Azithromycin, Ceftriaxone, Ciprofloxacin, Nalidixic Acid, Pivmecillinam, and Trimethoprim-Sulfamethoxazole and defined as intermediate or resistant according to the most recent Clinical and Laboratory Standards Institute (CLSI) interpretive standards at the time of data analysis.
Cost per episode treated | 3 months
  Cost per episode treated will be calculated using the direct and indirect financial costs and total economic costs of illness per outpatient and inpatient episode of Shigella-associated diarrhea from the household and, separately, payer perspectives.
Death | 3 months
  Death: all cause mortality during follow-up among enrolled children.
Hospitalization | 3 months
  Hospitalization will be defined as an overnight stay (child was on the ward from at least 12am to 6am) that occurs during follow-up among enrolled children
Persistent diarrhea (index episode) | 3 months
  Persistent diarrhea will be defined as 14 or more days of diarrhea (starting from the date at which the diarrhea first started (as opposed to date at presentation to an EFGH facility) and concluding at the last day of diarrhea prior to the two consecutive diarrhea-free days concluding the episode.
Diarrhea/dysentery recurrence | 3 months
  Diarrhea/dysentery recurrence will be defined as new diarrhea/dysentery episodes (>48 hours after a diarrhea-free period).
Change in linear growth | 3 months
  Change in mean length/height-for-age z-score (∆LAZ/∆HAZ) from enrollment to 3 months. The 2006 World Health Organization (WHO) reference population will be used to calculate HAZ from the average of two repeated length/height (cm) measures per child per time point

CONTACTS AND LOCATIONS:
Overall Officials: Patricia B Pavlinac, PhD, Principal Investigator — University of Washington
Locations (33):
- Bangladesh (5):
  - Dhaka Medical College Hospital, Dhaka
  - EFGH Field Clinic, Dhaka
  - icddr,b Dhaka Hospital, Dhaka
  - Mugda Medical College Hospital, Dhaka
  - Sir Salimullah Medical College Hospital, Dhaka
- Kenya (9):
  - Abidha Health Center, Siaya
  - Akala Health Center, Siaya
  - Bar Agulu Health Center, Siaya
  - Dienya Health Centre, Siaya
  - Lwak Mission Hospital, Siaya
  - Ongielo Health Centre, Siaya
  - Siaya County Referral Hospital, Siaya
  - Ting Wangi Health Center, Siaya
  - Wagai Health Center, Siaya
- Ndirande Health Centre, Blantyre, Malawi
- Mali (4):
  - Asacodjeneka Cscom, Bamako
  - Asacodjip Cscom, Bamako
  - Banconi CSCOM (ASACOBA), Bamako
  - CSREF Commune 1, Bamako
- Pakistan (6):
  - Abbasi Shaheed Hospital, Karachi
  - Ali Akbar Shah Center, Karachi
  - Bhains colony AKU site, Karachi
  - Khidmat e Alam Medical Centre, Karachi
  - Sindh Government Hospital, Ibrahim Hyderi, Karachi
  - Sindh Government Hospital, Korangi, Karachi
- Peru (6):
  - America Health Post, Iquitos, Maynas
  - Hospital de Apoloyo, Iquitos, Maynas
  - Modelo Health Post, Iquitos, Maynas
  - Progreso Health Post, Iquitos, Maynas
  - San Juan Health Post, Iquitos, Maynas
  - Santo Tomas Health Post, Iquitos, Maynas
- The Gambia (2):
  - Basse Hospital, Basse Santa Su, Upper River Division
  - Gambisara Health Centre (HC), Basse Santa Su, Upper River Division

IPD SHARING:
Plan to Share IPD: Yes
The publicly available analytic de-identified datasets corresponding to each specific aim, along with corresponding analytic code in Stata or R, will be posted to Dataverse, which is a publicly available data repository. Data requests for data not included in the publicly available analytic datasets corresponding to each aim will be managed by the University of Washington and relevant EFGH site investigators.
Supporting Information: Analytic Code

REFERENCES:
- [Background] Rogawski McQuade ET, Shaheen F, Kabir F, Rizvi A, Platts-Mills JA, Aziz F, Kalam A, Qureshi S, Elwood S, Liu J, Lima AAM, Kang G, Bessong P, Samie A, Haque R, Mduma ER, Kosek MN, Shrestha S, Leite JP, Bodhidatta L, Page N, Kiwelu I, Shakoor S, Turab A, Soofi SB, Ahmed T, Houpt ER, Bhutta Z, Iqbal NT. Epidemiology of Shigella infections and diarrhea in the first two years of life using culture-independent diagnostics in 8 low-resource settings. PLoS Negl Trop Dis. 2020 Aug 17;14(8):e0008536. doi: 10.1371/journal.pntd.0008536. eCollection 2020 Aug. PMID 32804926
- [Background] Kotloff KL, Nataro JP, Blackwelder WC, Nasrin D, Farag TH, Panchalingam S, Wu Y, Sow SO, Sur D, Breiman RF, Faruque AS, Zaidi AK, Saha D, Alonso PL, Tamboura B, Sanogo D, Onwuchekwa U, Manna B, Ramamurthy T, Kanungo S, Ochieng JB, Omore R, Oundo JO, Hossain A, Das SK, Ahmed S, Qureshi S, Quadri F, Adegbola RA, Antonio M, Hossain MJ, Akinsola A, Mandomando I, Nhampossa T, Acacio S, Biswas K, O'Reilly CE, Mintz ED, Berkeley LY, Muhsen K, Sommerfelt H, Robins-Browne RM, Levine MM. Burden and aetiology of diarrhoeal disease in infants and young children in developing countries (the Global Enteric Multicenter Study, GEMS): a prospective, case-control study. Lancet. 2013 Jul 20;382(9888):209-22. doi: 10.1016/S0140-6736(13)60844-2. Epub 2013 May 14. PMID 23680352
- [Background] Liu J, Platts-Mills JA, Juma J, Kabir F, Nkeze J, Okoi C, Operario DJ, Uddin J, Ahmed S, Alonso PL, Antonio M, Becker SM, Blackwelder WC, Breiman RF, Faruque AS, Fields B, Gratz J, Haque R, Hossain A, Hossain MJ, Jarju S, Qamar F, Iqbal NT, Kwambana B, Mandomando I, McMurry TL, Ochieng C, Ochieng JB, Ochieng M, Onyango C, Panchalingam S, Kalam A, Aziz F, Qureshi S, Ramamurthy T, Roberts JH, Saha D, Sow SO, Stroup SE, Sur D, Tamboura B, Taniuchi M, Tennant SM, Toema D, Wu Y, Zaidi A, Nataro JP, Kotloff KL, Levine MM, Houpt ER. Use of quantitative molecular diagnostic methods to identify causes of diarrhoea in children: a reanalysis of the GEMS case-control study. Lancet. 2016 Sep 24;388(10051):1291-301. doi: 10.1016/S0140-6736(16)31529-X. PMID 27673470
- [Background] Pavlinac PB, Rogawski McQuade ET, Platts-Mills JA, Kotloff KL, Deal C, Giersing BK, Isbrucker RA, Kang G, Ma LF, MacLennan CA, Patriarca P, Steele D, Vannice KS. Pivotal Shigella Vaccine Efficacy Trials-Study Design Considerations from a Shigella Vaccine Trial Design Working Group. Vaccines (Basel). 2022 Mar 22;10(4):489. doi: 10.3390/vaccines10040489. PMID 35455238
- [Background] Kasumba IN, Badji H, Powell H, Hossain MJ, Omore R, Sow SO, Verani JR, Platts-Mills JA, Widdowson MA, Zaman SMA, Jones J, Sen S, Permala-Booth J, Nasrin S, Roose A, Nasrin D, Ochieng JB, Juma J, Doh S, Jones JCM, Antonio M, Awuor AO, Sugerman CE, Watson N, Focht C, Liu J, Houpt E, Kotloff KL, Tennant SM. Shigella in Africa: New Insights From the Vaccine Impact on Diarrhea in Africa (VIDA) Study. Clin Infect Dis. 2023 Apr 19;76(76 Suppl1):S66-S76. doi: 10.1093/cid/ciac969. PMID 37074444
- [Background] von Seidlein L, Kim DR, Ali M, Lee H, Wang X, Thiem VD, Canh DG, Chaicumpa W, Agtini MD, Hossain A, Bhutta ZA, Mason C, Sethabutr O, Talukder K, Nair GB, Deen JL, Kotloff K, Clemens J. A multicentre study of Shigella diarrhoea in six Asian countries: disease burden, clinical manifestations, and microbiology. PLoS Med. 2006 Sep;3(9):e353. doi: 10.1371/journal.pmed.0030353. PMID 16968124

DOCUMENTS (2):
  • Statistical Analysis Plan (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT06047821/SAP_004.pdf
  • Informed Consent Form (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT06047821/ICF_002.pdf